CLINICAL TRIAL: NCT02592603
Title: Endocuff-assisted vs. Standard Colonoscopy for Surveillance of Serrated Polyposis Syndrome: A Randomized Controlled Trial
Brief Title: Endocuff for Surveillance of Serrated Polyposis Syndrome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital Clinic of Barcelona (Other)
Collaborators: Fundacion Clinic per a la Recerca Biomédica (Other)
Responsible Party: Principal Investigator, María Pellisé, MD. PhD. Consultant, Hospital Clinic of Barcelona
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: HCB/2015/0803
Record Dates: First submitted 2015-10-29; First posted 2015-10-30 (Estimated); Last update posted 2017-08-04 (Actual); Status verified 2017-08

CONDITIONS: Polyposis
Keywords: Serrated lesions; Surveillance; Colorectal cancer; Endocuff; Sessile serrated adenoma; Colonoscopy
MeSH Terms: conditions — Colorectal Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Endocuff-assisted Colonoscopy (Active Comparator): Endocuff-assisted Colonoscopy with the ARC Endocuff-vision® attached at the distal tip of the scope.
  Interventions: Device: Endocuff-assisted Colonoscopy
- Standard Colonoscopy (No Intervention): Standard Colonoscopy without any additional device

INTERVENTIONS:
Device: Endocuff-assisted Colonoscopy — Colonic examination with Endocuff-assisted Colonoscopy
  Other Names: ECC
  Arms: Endocuff-assisted Colonoscopy

SUMMARY:
Serrated Polyposis Syndrome (SPS) is a high-risk condition for colorectal cancer (CRC). SPS patients have a cumulative CRC risk of 1.9% in 5 years despite a strict endoscopic surveillance in specialized centers. Proximal serrated lesions are endoscopically challenging to detect due to their unremarkable morphology. Endocuff is a novel device comprised of a cap with a row of finger-like projections with a unique dynamic shape that help to flatten mucosal folds during withdrawal of the instrument in order to improve detection of lesions. Recent studies have reported an increase of detection rate and mean per patient of adenomas with Endocuff-assisted Colonoscopy compared with Standard Colonoscopy. The purpose of this study is to assess the usefulness of Endocuff-assisted Colonoscopy to detect serrated lesions in SPS patients undergoing surveillance compared to Standard Colonoscopy in a randomized fashion

DETAILED DESCRIPTION:
According to own data and similarly to previous published studies, patients diagnosed of Serrated Polyposis Syndrome undergoing annual surveillance after clearance of all serrated lesions ≥ 5mm, have a mean of 5 serrated lesions per patient at follow-up colonoscopies. The study was powered to establish a 25% significant increase in the mean of serrated lesions per patient in the Endocuff-assisted colonoscopy group. Accepting an alpha risk of 0.05, a beta risk of 0.2 and a loss rate of 10% in a bilateral contrast, a sample size of 124 patients (62 in each arm) are required to achieve statistic significance.

ELIGIBILITY:
Inclusion Criteria:

-Adults with diagnosis of Serrated Polyposis Syndrome undergoing surveillance colonoscopies after clearance of all lesions >=5mm

Exclusion Criteria:

* Patients with known strictures
* Partial or total colonic resection
* Acute diverticulitis
* Concomitant inflammatory bowel disease
* Suspected or proven lower gastrointestinal bleeding
* Non-correctable coagulopathy or anticoagulant/clopidogrel therapy during procedure
* Inability to sign informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 125 (Actual)
Dates: Start 2015-10; Primary Completion 2017-07 (Actual); Study Completion 2017-07 (Actual)

PRIMARY OUTCOMES:
Number of serrated lesions >=5mm | one year
  Number of serrated lesions >=5mm detected in each arm

SECONDARY OUTCOMES:
Number of total polyps | one year
  Number of total polyps in each arm
Number of serrated lesions >=10mm | one year
  Number of serrated lesions >=10mm detected in each arm
Number of serrated lesions with displasia | one year
  Number of serrated lesions with displasia in each arm
Number of adenomas | one year
  Number of adenomas in each arm
Number of advanced adenomas | one year
  Number of advanced adenomas in each arm
Number of flat lesions | one year
  Number of flat lesions in each arm
Number of flat lesions in right colon | one year
  Number of flat lesions in right colon in each arm
Withdrawal time | 30 minutes
  Extubation time from the cecum to scope removal from the anus, with exception of time taken for any therapeutic intervention
Total procedure time | 30 minutes
  Starting with endoscope insertion and withdrawal time including therapeutic interventions
Proportion of major adverse events | Two weeks
  Colonic perforation or clinically significant bleeding
Proportion of minor adverse events | Two weeks
  Superficial mucosal erosions in the colonic mucosa, abdominal pain and bloating

CONTACTS AND LOCATIONS:
Overall Officials: María Pellisé, MD. PhD, Principal Investigator — Hospital Clinic of Barcelona
Locations (1):
- María Pellisé. MD. PhD., Barcelona, Spain

REFERENCES:
- [Background] Carballal S, Rodriguez-Alcalde D, Moreira L, Hernandez L, Rodriguez L, Rodriguez-Moranta F, Gonzalo V, Bujanda L, Bessa X, Poves C, Cubiella J, Castro I, Gonzalez M, Moya E, Oquinena S, Clofent J, Quintero E, Esteban P, Pinol V, Fernandez FJ, Jover R, Cid L, Lopez-Ceron M, Cuatrecasas M, Lopez-Vicente J, Leoz ML, Rivero-Sanchez L, Castells A, Pellise M, Balaguer F; Gastrointestinal Oncology Group of the Spanish Gastroenterological Association. Colorectal cancer risk factors in patients with serrated polyposis syndrome: a large multicentre study. Gut. 2016 Nov;65(11):1829-1837. doi: 10.1136/gutjnl-2015-309647. Epub 2015 Aug 11. PMID 26264224
- [Background] Biecker E, Floer M, Heinecke A, Strobel P, Bohme R, Schepke M, Meister T. Novel endocuff-assisted colonoscopy significantly increases the polyp detection rate: a randomized controlled trial. J Clin Gastroenterol. 2015 May-Jun;49(5):413-8. doi: 10.1097/MCG.0000000000000166. PMID 24921209
- [Background] Floer M, Biecker E, Fitzlaff R, Roming H, Ameis D, Heinecke A, Kunsch S, Ellenrieder V, Strobel P, Schepke M, Meister T. Higher adenoma detection rates with endocuff-assisted colonoscopy - a randomized controlled multicenter trial. PLoS One. 2014 Dec 3;9(12):e114267. doi: 10.1371/journal.pone.0114267. eCollection 2014. PMID 25470133
- [Background] Sawatzki M, Meyenberger C, Marbet UA, Haarer J, Frei R. Prospective Swiss pilot study of Endocuff-assisted colonoscopy in a screening population. Endosc Int Open. 2015 Jun;3(3):E236-9. doi: 10.1055/s-0034-1391418. Epub 2015 Feb 27. PMID 26171436
- [Derived] Rivero-Sanchez L, Lopez Vicente J, Hernandez Villalba L, Puig I, Arnau-Collell C, Moreno L, Diaz M, Rodriguez de Miguel C, Ocana T, Moreira L, Cuatrecasas M, Carballal S, Sanchez A, Ortiz O, Llach J, Balaguer F, Pellise M; EndoCAR group from the Spanish Gastroenterology Association and the Spanish Society of Digestive Endoscopy. Endocuff-assisted colonoscopy for surveillance of serrated polyposis syndrome: a multicenter randomized controlled trial. Endoscopy. 2019 Jul;51(7):637-645. doi: 10.1055/a-0925-4956. Epub 2019 Jun 7. PMID 31174224